CLINICAL TRIAL: NCT04938661
Title: Improving Cardiac Rehabilitation Outcomes Through Mobile Case Management (iCARE)
Acronym: iCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Thomas P. Olson, M.S., Ph.D., Associate Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-002258; R01NR018832 (NIH)
Record Dates: First submitted 2021-05-14; First posted 2021-06-24 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Acute Myocardial Infarction; Acute Coronary Syndrome; Stable Angina Pectoris; Percutaneous Coronary Intervention; Heart Failure
Keywords: Cardiac Rehabilitation
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Stable; Heart Failure | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Center-Based Cardiac Rehab (CON) (Active Comparator): Participants will be prescribed 36 sessions of center-based CR. This includes supervised exercise sessions, cooking demonstrations, didactic lectures, video presentations, group support, and stress management education. During sessions, participants have direct access to the medical director, case manager, registered nurse, exercise physiologist, and stress management specialists.
  Interventions: Other: Center-Based Cardiac Rehab
- Conventional Center-Based Cardiac Rehab + mHealth (CON+) (Active Comparator): Participants will be prescribed 36 sessions of center-based CR as noted above. In addition, participants will be provided access to the mHealth platform which provides "e-Learning modules" with factsheets, videos, quizzes, and questionnaires (coinciding with activities being conducted during the CON program), a Social Network Module will allow patients to communicate via secure network with other patients who are part of their invited network. The Social Network Module also allows for secure two-way interaction with healthcare providers in the event that patients are experiencing signs or symptoms suggestive of worsening condition. This platform also contains a Personal Health Record Module allowing patients to upload, archive, and retrieve personal health data (e.g. fitness tracker data, heart rate monitor data, blood pressure recordings, etc.) and record vital signs, symptoms, treatments, and medical history.
  Interventions: Other: Center-Based Cardiac Rehab; Other: mHealth
- Home-Based Cardiac Rehab + mHealth (HOM+) (Active Comparator): Participants will be provided paper copies of educational content at the time of event/discharge. In addition, these participants will be provided access to the same mHealth platform as the CON+ group. Participants in this group will be encouraged to exercise three days per week while also completing the additional questionnaires and educational content provided by the mHealth platform in accordance with the CR program. Participation will be tracked using web/internet analytics.
  Interventions: Other: mHealth; Other: Home-Based Cardiac Rehab

INTERVENTIONS:
Other: Center-Based Cardiac Rehab — 36 center-Based Cardiac Rehab Sessions
  Arms: Conventional Center-Based Cardiac Rehab (CON); Conventional Center-Based Cardiac Rehab + mHealth (CON+)
Other: mHealth — Mobile Health Platform
  Arms: Conventional Center-Based Cardiac Rehab + mHealth (CON+); Home-Based Cardiac Rehab + mHealth (HOM+)
Other: Home-Based Cardiac Rehab — Encouraged to exercise 3 times per week at home
  Arms: Home-Based Cardiac Rehab + mHealth (HOM+)

SUMMARY:
The purpose of this research is to find out if doing cardiac rehab at home, or a mix of cardiac rehab at home and in the clinic, is as effective as coming in to the clinic for cardiac rehab.

DETAILED DESCRIPTION:
To address our specific aims we will use a single-center, prospective, three-arm, parallel group, randomized controlled trial design. At the time of identification of eligibility for participation, patients will be randomized to one of three arms (1:1:1 ratio): Arm 1 consists of patients randomized to conventional cardiac rehab only, Arm 2 consists of patients randomized to conventional cardiac rehab with the addition of the mHealth platform, and Arm 3 consists of patients randomized to remote case management using the mHealth platform only. Clinical metrics will include traditional cardiovascular risk factors with additional tracking of service utilization and adherence, and quality of life. Measures will be made at baseline (pre-intervention) and ~3-months (coinciding with completion of conventional CR). Additional follow-up will occur at 12 months post CR entry. Randomization to study arms will be done with a multidimensional dynamic allocation algorithm, minimizing imbalances in age, sex, body mass index, and race across study arms.

ELIGIBILITY:
Inclusion Criteria:

* Own or have reliable access to a smartphone or desktop computer with internet access
* Have an email address
* Patients who have a history of one of the following; acute myocardial infarction/acute coronary syndrome, stable angina pectoris, percutaneous coronary intervention, or heart failure.
* Patients who have undergone a surgical procedure which includes an indication for cardiac rehabilitation (coronary artery bypass surgery, heart valve repair/replacement, or heart transplant)

Exclusion Criteria:

* Patients referred to cardiac rehab with ventricular assist devices.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Functional Capacity | 3 Months
  VO2 peak
Number of participants who are re-hospitalized during the trial | 1 Year
  We will look at the number of patients who are hospitalized for any reason during the follow-up period

SECONDARY OUTCOMES:
Change in Body Weight | 3 Months
  body weight will be measured from pre to post intervention to see if weight decreases
Fasting Basic Lipid Panel | 3 Months
  All fasting blood chemistry measures will be conducted by standard clinical protocols in the Mayo Clinic laboratories. These measures will be conducted at the time of enrollment in the research program and during each of the two follow-up study visits.
Fasting Blood Glucose | 3 Months
  All fasting blood chemistry measures will be conducted by standard clinical protocols in the Mayo Clinic laboratories. These measures will be conducted at the time of enrollment in the research program and during each of the two follow-up study visits.
Fasting Hemoglobin | 3 Months
  All fasting blood chemistry measures will be conducted by standard clinical protocols in the Mayo Clinic laboratories. These measures will be conducted at the time of enrollment in the research program and during each of the two follow-up study visits.
Fasting Hemoglobin A1C | 3 Months
  All fasting blood chemistry measures will be conducted by standard clinical protocols in the Mayo Clinic laboratories. These measures will be conducted at the time of enrollment in the research program and during each of the two follow-up study visits.
6 Minute Walk Test | 3 Months
  exercise capacity
Self-Reported Physical Activity | 3 Months
  assessed via IPAQ questionnaire
Self-Reported Physical Activity | 3 Months
  assessed via DASI questionnaire
Self-Reported Dietary Patterns | 3 Months
  obtained using a standard food frequency questionnaire
Self-Reported Quality of Life | 3 Months
  Assessed using PHQ-9
Self-Reported Quality of Life | 3 Months
  Assessed using Darmouth 9-item short-form health survey

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Olson, Ph.D., M.S., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2024-09-27): https://cdn.clinicaltrials.gov/large-docs/61/NCT04938661/ICF_000.pdf